CLINICAL TRIAL: NCT04506541
Title: The Effects Of Birth Kangaroo Care On Exclusively Breastfeeding And Baby's Growth And Development According To Attachment Theory
Brief Title: The Effects Of KC On Exclusively Breastfeeding And Baby's Growth And Development According To Attachment Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Buca Women Birth and Child Diseases Hospital (Unknown)
Responsible Party: Principal Investigator, Emine Serap Sarıcan, Principal Investigator, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kangaroo care at birth
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Breastfeeding, Exclusive; Growth Acceleration; Development, Infant; Attachment
Keywords: kangaroo care; growth; development; breastfeeding; maternal attachment
MeSH Terms: conditions — Breast Feeding | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo Care Group (Experimental): The pregnant women who were in the kangaroo care group of the study and who were 36-38 weeks of gestation were given 20 minutes of kangaroo care and breastfeeding training by the researcher. A video about "kangaroo care and breastfeeding" was sent to pregnant women to remind them two weeks after the training. Kangaroo care application started in the first minute after giving birth in mothers who were in the kangaroo care group and came to the delivery room. In the first, third, sixth, and ninth months after the discharge of the mothers who started applying kangaroo care, kangaroo care application status, breastfeeding status, baby's growth, and development status were evaluated. In each follow-up, the baby's height, weight, and head circumference were measured with a standard measuring tool.
  Interventions: Other: Kangaroo Care
- Control Group (No Intervention): The pregnant women in the control group were not trained other than breastfeeding training given in the hospital. In the maternity room, routine care practices were performed after delivery of the pregnant women. As in mothers in the kangaroo care group, in the first, third, sixth, and ninth months after the discharge of mothers, kangaroo care application situations, breastfeeding conditions, growth, and development of the baby were evaluated.

INTERVENTIONS:
Other: Kangaroo Care — Kangaroo care application started in the first minute after giving birth in mothers who were in the kangaroo care group and came to the delivery room.
  Arms: Kangaroo Care Group

SUMMARY:
Kangaroo care is a developmental care method determined to improve the quality of life of premature babies. When the benefits of kangaroo care on development and feeding with breast milk on premature babies are considered, term babies should also receive kangaroo care, and kangaroo care should be started immediately after birth. In this research, the authors aimed to investigate the effect of kangaroo care at birth on breast milk only feeding status and infant growth and development according to attachment theory. This is a randomized controlled, experimental, prospective study. The sample of the study consisted of pregnant women between 36-38 gestational weeks, who referred to the pregnant outpatient clinic of Buca Maternity and Children Hospital between March 2017 and February 2019 (n: 132). Pregnant women in the intervention group received "kangaroo care and breastfeeding training," and their babies were given kangaroo care at birth. Routine care was given to the mothers and their babies in the control group. Maternal attachment levels of mothers in both groups after birth and infants' breastfeeding only status and infant growth and development in the first, third, sixth, and ninth months were evaluated.

DETAILED DESCRIPTION:
The research is a randomized controlled, experimental, prospective study conducted to examine the effect of kangaroo care at birth on feeding with breast milk only and nutritional status and growth-development of the baby according to attachment theory. The research was carried out at the Republic of Turkey, Ministry of Health, Izmir Provincial Health Directorate, Buca Women Birth and Child Diseases Hospital. The population of the study consisted of all pregnant women who were between 36-38 weeks of gestation and referred to the pregnant outpatient clinic between March 2017 and February 2019 (N.8079).Power analysis was carried out to determine the sample group that would represent the population in the research. In the power analysis, the sample was determined by evaluating the reference studies related to the feeding rate of only with breast milk in the first nine months, and the expected growth development level in the first nine months, which were the dependent variables of the research. For the first nine months, the 2.4% value stated in TNSA 2013 regarding feeding with breast milk rate was taken as reference (TNSA, 2013). Studies of Çelik et al. (2014) were taken as reference for the evaluation of growth and development. The number of samples to be taken for each group was determined as a result of the power analysis made according to these values. As a result of the evaluation made with power analysis, the expected effect factor with growth and development was calculated as two-times. Accordingly, it was determined that 48 samples should be taken for each group. Forecasting that data loss may occur in multi-monitoring studies, more than 10% of the sufficient sample size was included in the study (n: 214). The sample of the study consisted of pregnant women who applied to the Ministry of Health, Izmir Provincial Health Directorate, Buca Women Birth and Child Diseases Hospital pregnant outpatient clinic between March 2017 and February 2019, who were between 36-38 weeks of gestation and who met the inclusion criteria (n:132). After determining the sample number of the research, it was decided to make randomization according to the last numbers of the pregnant women's protocol numbers, and to which group the odd and even numbers would be included was determined by the method of a draw. As a result of the draw, the last digit of the protocol number ending with an odd number was included in the control group, the last digit of the protocol number, ending with an even number, was included in the intervention group

ELIGIBILITY:
The inclusion criteria

* 36-38 gestational weeks,
* giving birth at 37 weeks or above,
* single and live fetus,
* having no obstacle for applying kangaroo care,
* accepting kangaroo care implementation,
* no need for intervention of newborn,
* no need of newborn to be referred to the neonatal intensive care unit,
* being able to communicate with the pregnant woman,
* having a cesarean section with spinal or epidural anesthesia.

Exclusion criteria

* being accepted to the delivery room with urgent delivery,
* mothers who did not want to apply kangaroo care,
* mothers who had mental disorders which could harm the baby or self such as postpartum depression,
* the delivery was performed under general anesthesia for pregnant women who had a cesarean delivery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
breastfeeding conditions | from birth to the ninth month
  Baby's time to start sucking: how many minutes in the first half hour it starts to suck Absorption time: How many minutes it absorbs in the first half hour
  o Breastfeeding status only: Breastfeeding time of the mother's baby only until the end of the research by using Kangaroo Care and Breastmilk Intake Status Inspection Form. The form was developed by the researcher to monitor and control how long the mother implemented the kangaroo care, the time baby started breastfeeding, the duration of breastfeeding, and the changes in the baby's body weight
baby's weight | from birth to the ninth month
  the weight of the baby was evaluated in grams and was measured with a standard measuring tool.
baby's height | from birth to the ninth month
  the height of the baby was evaluated in centimeter and was measured with a standard measuring tool.
baby's head circumferecne | from birth to the ninth month
  the head circumference of the baby was evaluated in centimeter and was measured with a standard measuring tool.
baby's development | from birth to the ninth month
  Baby's first, third, sixth and ninth month developmental status by using Guide to Monitoring and Supporting Development. There is no scoring in the development monitoring and supporting guide. In the study, the developmental status of the babies was categorized as "behind by month," "normal by month," and "ahead by month.
maternal attachment | from birth to the ninth month
  Attactment level between mother and baby at postpartum first, third, sixth and ninth months by using Maternal Attachment Scale. The scale consists of 26 items in a four-point Likert type. The minimum score that can be obtained from the scale is 26, the maximum score is 104, and the height of the score indicates that the bond between the mother and the baby is high The Cronbach's alpha value of the scale was determined as 0.87 in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia GENÇ, Principal Investigator — Ege University
Locations (1):
- Ege University, Bornova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No